CLINICAL TRIAL: NCT03248050
Title: Evaluating an Intervention to Increase Use of Call Centre Support for Self-managed Medical Abortion, and the Effectiveness of Call Centre Support for Correct Use of Medical Abortion: A Cluster Randomised-controlled Trial With Nested Observational Study
Brief Title: Evaluating an Intervention to Increase Use of Call Centre Support for Self-managed Medical Abortion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Marie Stopes International (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 011-17
Record Dates: First submitted 2017-06-23; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Abortion, Drug-Induced; Pharmacies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention pharmacy (Experimental): Pharmacies in the intervention group will receive training, materials, and monitoring visits to encourage them to inform women who buy mifepristone + misoprostol or misoprostol alone to call the MSZ call centre for advice on how to use the pills before they take them.
  Interventions: Behavioral: Pharmacy encouraged to promote call centre use to clients
- Control pharmacy (No Intervention)

INTERVENTIONS:
Behavioral: Pharmacy encouraged to promote call centre use to clients — The details of the intervention will be finalised following an intervention design workshop. The main components will be: Provision of materials with the MSZ call centre number on for pharmacy workers to give women buying MA medications to call the number for free, confidential advice on how to use the pills before they take them; incentives; monthly monitoring visits.
  Arms: Intervention pharmacy

SUMMARY:
Self-management of medical abortion (MA) pills purchased from pharmacies is considered to be one of the reasons behind falling morbidity and mortality from unsafe abortion in recent years. While pharmacy workers commonly sell MA medications over the counter, they have inadequate knowledge about how women should take the medications and their potential complications, and do not offer adequate information and counselling to women buying the drugs. This study aims to evaluate if a pharmacy-based intervention to promote use of a support hotline (Marie Stopes Zambia (MSZ) call centre) among MA purchasers can increase use of the call centre, and to assess whether correct MA use and acceptability of self- administered MA is higher among MA users who contact the call centre than those who self-administer MA without call centre support.

DETAILED DESCRIPTION:
Self-management of medical abortion (MA) pills purchased from pharmacies is considered to be one of the reasons behind falling morbidity and mortality from unsafe abortion in recent years. While pharmacy workers commonly sell MA medications over the counter, they have inadequate knowledge about how women should take the medications and their potential complications, and do not offer adequate information and counselling to women buying the drugs.

This study aims to evaluate if a pharmacy-based intervention to promote use of a support hotline (Marie Stopes Zambia (MSZ) call centre) among MA purchasers can increase use of the call centre, and to assess whether correct MA use and acceptability of self- administered MA is higher among MA users who contact the call centre than those who self-administer MA without call centre support.

The objectives of the study are:

1. To evaluate whether a pharmacy-based intervention to promote the MSZ call centre increases contact with the call centre among women purchasing the combination regimen or misoprostol alone from pharmacies for MA.
2. To evaluate whether a pharmacy-based intervention to promote the MSZ call centre can increase the proportion of pharmacy workers encouraging mystery clients purchasing the combination regimen or misoprostol-only to use the MSZ call centre.
3. To assess the reasons for use and non-use of the call centre advice line among women purchasing MA from pharmacies
4. To investigate whether correct MA regimen use and acceptability of self-administered MA are higher among those women who call the call centre, compared to those who self-administer MA without any call centre support.

The details of the programme intervention will be finalised following an intervention design workshop but the main components will be as follows:

* Provide pharmacy workers with either paper pill bags, cards to put in existing pill bags, or stickers to put on pill packaging, which have the MSZ call centre number printed on them, along with instructions to ring the hotline for free, confidential advice about reproductive health issues.
* Train all pharmacy workers at the pharmacy through one-on-one detailing visits to encourage all clients buying misoprostol (any brand) or the mifepristone-misoprostol combined regimen (any brand) to call the number for free, confidential advice on how to use the pills before they take them.
* Incentivise pharmacy workers to encourage women to phone the call centre.s.
* Monthly monitoring visits to remind pharmacy workers to encourage women to phone the free, confidential phone number (in person or remotely through phone calls).

Women who call the call centre will receive advice on how to take the MA medications. Call centre staff will have a script detailing essential information on MA and answers to possible client questions.

To evaluate this intervention, a two arm, single group, superiority, multicentre, cluster randomised controlled trial with a nested observational study will be conducted at 26 pharmacies in Lusaka, Zambia. A randomised trial design will be used to assess the effectiveness of the pharmacy-based intervention in increasing use of the call centre. As it is not possible to randomly assign women to actually use the call centre and use will be largely based on self-selection, the nested observational study will then compare the experience of women who use and do not use the call centre.

Data collection will include:

1. Structured interviews with women using medications purchased from pharmacies to assess call centre use, MA regimen used, and experience of self-administering MA (impact evaluation and nested-observational study), and
2. Mystery client surveys to assess pharmacy practice (process evaluation).
3. Qualitative analysis of a sample of call recordings (process evaluation).
4. Costing analysis of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Pharmacies:

* Located in Lusaka
* Supplied with MSZ's Mariprist combination regimen product
* Selling > 10 products per month
* Pharmacy owner and at least one pharmacy worker is willing to participate

MA users:

* Women using combination regimen or misoprostol-alone for MA, purchased from study pharmacies during the study period
* Purchased medication by themselves or by a proxy purchaser
* Have access to a mobile phone and are willing to be followed up by phone with questions about her abortion at 14 and 60 days after taking the first drug
* Aged 18 and over
* Certain of the date of their last menstrual period (LMP) and have gestational age less than 9 weeks (calculated from LMP)
* Have a confirmed pregnancy (self-reported positive urine pregnancy test)
* Willing and able to give informed consent

Mystery clients:

* Aged 18 and over
* Female
* Not pregnant
* Literate
* Pro-choice
* Not current or former employees of pharmacies
* Not related to current or former employees of pharmacies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1359 (Estimated)
Dates: Start 2017-10-15 (Estimated); Primary Completion 2018-04-15 (Estimated); Study Completion 2018-06-15 (Estimated)

PRIMARY OUTCOMES:
Self-reported use of call centre in past two weeks | Day 14 after taking the first pill
  Participant called MSZ call centre after purchasing the medication.
Self-reported use of a correct regimen of MA | Day 14 after taking the first pill
  Use of a correct regimen of mifepristone-misoprostol: 200mg mifepristone (oral administration) followed by single dose of 800mcg misoprostol (vaginal, buccal or sublingually), or 400mcg misoprostol orally if under 7 weeks gestation, after a 24-48 hour interval. Use of a correct regimen of misoprostol only: 800mcg of misoprostol vaginally or sublingually, with subsequent doses of 800 mcg every 3 hours up to 3 doses
Self-reported satisfaction with self-administration of MA | Day 14 after taking the first pill
  Satisfaction with the overall process, would recommend to a friend who needed an abortion, would use the same method again if needed an abortion again, feeling adequately prepared for various aspects of the medical abortion process.

SECONDARY OUTCOMES:
Cost of intervention per unit of call centre use | Day 14 after taking first pill
  Increased unit cost of intervention per increased unit of call centre use.
Self-reported abortion completion rate | Day 14 and day 60 after taking first pill
  Proportion of women self-reporting that at day 60, they are no longer pregnant(due to self-reported negative result of a urine pregnancy test, self-reported expulsion of pregnancy, self-reported return to regular menstrual cycles, self-reported disappearance of pregnancy symptoms or all of the above), without recourse to a repeat procedure (surgical or medical).
Self-reported uptake of post-abortion family planning | Day 14 after taking first pill
  Uptake of a post abortion contraceptive: the respondent is using tubal ligation, intrauterine device, implant, injectable, or oral contraceptive pill at day 14 that she has started to use since taking the MA product.
Self-reported complication rate | Day 14 after taking first pill
  Hemorrhage requiring a blood transfusion or uterine aspiration, serious infection from the abortion needing IV antibiotics and undiagnosed (at the time of MA administration) ectopic pregnancy needing surgery or other treatment, a continuing pregnancy needing an uterine aspiration, an incomplete abortion needing uterine aspiration or further medication, severe allergic reaction, severe vomiting or diarrhea and admission to a health facility for any of the above.

OTHER OUTCOMES:
Proportion of pharmacy workers encouraging mystery clients to use the MSZ call centre number | Within 4 weeks of intervention starting
  During mystery client visit, pharmacy worker verbally mentions the MSZ call centre to the mystery client.
Proportion of mystery clients that receives study materials with call centre phone number on. | Within 4 weeks of intervention starting
  During the mystery client visit, pharmacy worker provides the mystery client with the study intervention materials that have the call centre number on.
Reasons for use and non-use of the call centre advice line | Day 14 after taking first pill
  MA users' self-reported reasons for calling or not calling the call centre.

IPD SHARING:
Plan to Share IPD: Undecided